CLINICAL TRIAL: NCT00239850
Title: Morbid Obesity: Effects of Conservative Treatments and Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2005.33; NSD12820 (Other: NSD); 05/3344TSP (Other: TSP)
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Morbid Obesity
Keywords: obesity; lifestyle; treatment; Complications; endocrine changes; Lipids; C18.654.726.500.495
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: lifestyle changes

SUMMARY:
The purpose of this study is to evaluate the effects of conservative treatments of obesity with surgery (gastric bypass).

DETAILED DESCRIPTION:
The aim of this study is to evaluate 3 different treatments of obesity with gastric bypass. Two groups will be treated in different clinics and 1 group will be treated at our outpatient clinic. Sixty patients will participate in each group. Behavioural changes and weight loss over 4-5 years will be followed. We will also analyse changes in hormones, mental status, sexual behaviour, effect of training and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 40 or BMI > 35 with complications

Exclusion Criteria:

* Unstable atherosclerotic disease
* Psychologically unstable
* Unable to participate in the training program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
weight reduction
quality of life

SECONDARY OUTCOMES:
reduction in obesity complications

CONTACTS AND LOCATIONS:
Overall Officials: Baard Kulseng, PhD, MD, Principal Investigator — St. Olavs Hospital, Trondheim; Ronald Mårvik, PhD, MD, Principal Investigator — St. Olavs Hospital, Trondheim
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Martins C, Strommen M, Stavne OA, Nossum R, Marvik R, Kulseng B. Bariatric surgery versus lifestyle interventions for morbid obesity--changes in body weight, risk factors and comorbidities at 1 year. Obes Surg. 2011 Jul;21(7):841-9. doi: 10.1007/s11695-010-0131-1. PMID 20379796
- [Result] Ovrebo B, Strommen M, Kulseng B, Martins C. Bariatric surgery versus lifestyle interventions for severe obesity: 5-year changes in body weight, risk factors and comorbidities. Clin Obes. 2017 Jun;7(3):183-190. doi: 10.1111/cob.12190. Epub 2017 Mar 20. PMID 28320081